CLINICAL TRIAL: NCT06802471
Title: Efficacy and Central Mechanism of Electroacupuncture for Medication Overuse Headache: a Multicenter Randomized Controlled Trial
Brief Title: Efficacy and Central Mechanisms of Electroacupuncture for Medication Overuse Headache
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, weiming wang, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-045-KY
Record Dates: First submitted 2025-01-21; First posted 2025-01-31 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Medication Overuse Headache; Electroacupuncture
MeSH Terms: conditions — Headache Disorders, Secondary | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- elecrtoacupuncture group (EA group) (Experimental): Participants will be treated by electroacupuncture. They will be treated 3 sessions a week for the first 6 weeks and 2 sessions a week (once every 2-3 days) for the next 6 weeks. The total course of treatment was 30 times for 12 weeks, each electroacupuncture treatment session for patients will be 30 minutes in duration. All the participants will be accepted usual care:
  Health education is provided in three aspects: lifestyle changes, behavioral therapies and MOH self-management.
  Basic treatment: Throughout the study period, patients could continue to use their previously overused symptomatic medications as usual. MOH patients are required not to change the type, single dose, or formulation of acute medications. However, they are allowed to increase or decrease the frequency or total amount of use based on their pain condition. Any use of new medications must be accurately documented.
  Interventions: Device: electroacupuncture
- Sham elecrtoacupuncture group (SEA group) (Sham Comparator): Participants will be treated by sham elecrtoacupuncture. They will be treated 3 sessions a week for the first 6 weeks and 2 sessions a week (once every 2-3 days) for the next 6 weeks. The total course of treatment was 30 times for 12 weeks, each electroacupuncture treatment session for patients will be 30 minutes in duration. All the participants will be accepted usual care:
  Health education is provided in three aspects: lifestyle changes, behavioral therapies and MOH self-management.
  Basic treatment: Throughout the study period, patients could continue to use their previously overused symptomatic medications as usual. MOH patients are required not to change the type, single dose, or formulation of acute medications. However, they are allowed to increase or decrease the frequency or total amount of use based on their pain condition. Any use of new medications must be accurately documented.
  Interventions: Device: Sham electroacupuncture
- Control group 1（CG 1） (No Intervention): Control group consisted of episodic migraine , they were matched to the MOH patient group by gender and age. Participants will undergo a clinical interview once a month, complete the headache diary assessment, have counseling and health education, and rescue medication if necessary. Health education is provided in three aspects: lifestyle changes, behavioral therapies and episodic migraine self-management.
  Participants will undergo brain MRI scans at baseline and at the end of week 12. Additionally, EA treatment and other interventions or treatments were not allowed throughout the 12-week study period.
- Control group 2（CG 2） (No Intervention): Control group 2 consisted of Healthy Volunteers , they were matched to the MOH patient group by gender and age.
  Participants will undergo brain MRI scans at baseline and at the end of week 12. Additionally, EA treatment and other interventions or treatments were not allowed throughout the 12-week study period.

INTERVENTIONS:
Device: electroacupuncture — The supine position, the local skin of the acupoints was routinely sterilized, and the selected acupoints were pasted with Acupuncture auxiliary device.
  The main acupuncture points are DU20, bilateral EX-HN5, ST8, GB20, GB20, LI4, LR3, ST40.
  Select compatible acupoints based on the patient's accompanying symptoms: 1.Discomfort in the neck: EX-B2 of Cervical 3-4; 2.Emotional anxiety, depression or sleep disorders: GV29, HT7; 3.Stomach or abdominal discomfort: CV12, ST25 and CV6.
  The disposable acupuncture needles and the electronic acupuncture treatment instrument SDZ-V nerve and muscle intimulator both manufactured by Suzhou Medical Appliance Factory Co., Ltd., China.The specifications of acupuncture needles are Φ0.30×25mm, Φ0.30×40mm, Φ0.30×50mm. The needles will be inserted into the skin of acupuncture points and manipulated manually by using the techniques such as lifting, thrusting, and twirling, until the internal compound sensation known as deqi.
  Arms: elecrtoacupuncture group (EA group)
Device: Sham electroacupuncture — The SEA group will use Hua Tuo brand disposable non-insertive sham control needles (Φ0.3mm×40mm) and the electronic acupuncture treatment instrument SDZ-V nerve and muscle intimulator both manufactured by Suzhou Medical Appliance Factory Co., Ltd., China. Sham points 1-2, 3-4, 5-6, and 7-8 are bilaterally located at the midpoints between the following pairs of acupoints: SP19 and EX-UE12, SP6 and LR5, EX-UE1 and HT1, and HT7 and SI8. sham LI4: Bilateral of midpoint between acupoint LI4 and LU9; sham LR3: Bilateral of midpoint between acupoint LR3 and ST44; sham ST40: Bilateral of midpoint between acupoint ST40 and GB35. Compatible acupoints: EX-B2 of Cervical 3-4 horizontal side by 0.5 cun; sham GV29: midpoint between acupoint GV29 and BL2. sham CV12: midpoint between acupoint CV12 and ST21; sham ST25: Bilateral of midpoint between acupoint ST25 and SP15; sham CV6: 3 cun lateral to the level of the CV6; The width of the interphalangeal joint of the patient's thumb was 1 "cun".
  Arms: Sham elecrtoacupuncture group (SEA group)

SUMMARY:
Acupuncture is commonly used for the prevention of migraine and tension-type headaches, and has been found to be effective in reducing both the frequency and severity of these conditions. However, studies on acupuncture for medication overuse headache (MOH) are limited, and current research has not been able to determine whether its efficacy is due to the actual therapeutic effects of acupuncture or psychological benefits. To address this issue, the investigators have designed a clinical trial to evaluate the efficacy of acupuncture for MOH. In addition, the investigators will explore the regulatory effects of electroacupuncture on central mechanisms in MOH and conduct multi-omics analysis.

DETAILED DESCRIPTION:
This is a multicenter, stratified, randomized, sham-controlled clinical trial. 120 eligible participants will be randomly allocated into electroacupuncture (EA), sham electroacupuncture (SEA), in a 1:1 ratio, which was divided into two phases

Phase 1 :

1. The EA group will receive 30 electroacupuncture treatments over an 12-week period, while the SEA group will receive sham electroacupuncture treatments with non-penetrating needling.

The two control groups are matched to the MOH patient group by gender and age for recruitment when the planned MOH patient enrollment was nearly 80% complete, and 20 patients in each group will be included, for a total of 40 patients.

Health education will be provided to participants in each group. The primary outcomes will be the changes of headache days per month from baseline after 12 weeks of treatment; The secondary outcomes will be as follows: The change from baseline in the number of headache days per month was also evaluated after 4 weeks of treatment, 8 weeks of treatment, 24 weeks of follow-up, and 36 weeks of follow-up; The proportion of responders, Headache Days per month, average daily headache time, headache Severity, average daily moderate-to-severe headache days, average daily moderate-to-severe headache time, Days with acute medication, Doses taken monthly, Severity of Dependence Scale, Headache Impact Test, EQOL-5D-5L, Hospital Anxiety and Depression Scale, Patients'expectation of the acupuncture efficacy, The Patient Global Impression of Change, The patient blinding assessment, Brain MRI Data Analysis and Multi-omics Analysis; The central randomization and data collection will be conducted by an electronic data management system.

Phase 2:

participants who adhere to the study protocol and complete the Week 36 follow-up will be considered to have completed the study. If the results of the first-phase trial demonstrate that electroacupuncture is superior to the control group, and the participants' willingness is confirmed, those willing to proceed will undergo the second-phase follow-up.

The second phase of follow-up was conducted at 1, 2, and 3 years after the end of treatment.These included whether the participant was lost to follow-up, headache diary (including headache frequency and medication use), recurrence of MOH, new comorbidities, and assessments using SDS, HIT-6, HADS, PGIC, and EQ-5D-5L.

ELIGIBILITY:
Inclusion Criteria for Patients with MOH:

* Meet the diagnostic criteria of MOH in ICHD-3;
* A history of migraine (according to ICHD-3 criteria)/tension headache (TTH) (according to ICHD-3 criteria) for ≥12 months before screening;
* Patients entered data from the electronic headache diary for at least 24 of the 28 days of the screening period (evidence of good adherence to the electronic headache diary);
* Prospectively collected data from the electronic headache diary during the screening period met the following criteria: 15 or more headache days per month; Regular overdose of acute or symptomatic headache medications meets the diagnostic criteria for MOH；
* Headache diagnosed before the age of 50 years;
* Patients had failed MOH withdrawal treatment (with medical documentation or specific physician confirmation of each treatment) on ≥1 occasions in the previous 3 years; Withdrawal treatment failure is defined as no significant reduction in headache frequency, duration and/or severity after withdrawal treatment; Or intolerable withdrawal reactions during withdrawal treatment; Or unable to quit treatment due to safety issues;
* Aged between 18 and 80 years old;
* Signed the informed consent and volunteered to participate in the study.
* Patients who met the above 8 criteria were included in this study.

Exclusion Criteria for Patients with MOH:

* Patients had a history or diagnosis of hypotensive headache, continuous hemiplegia, new daily persistent headache, or unusual migraine subtypes, such as hemiplegic migraine (sporadic and familial), ocular tension migraine, migraine with neurologic symptoms that were atypical of migraine aura (diplopia, altered consciousness, or prolonged duration). Other types of primary or secondary headache;
* The presence of clinically significant pain syndromes that may be confusing (e.g., fibromyalgia, chronic low back pain, complex regional pain syndrome); Acute or active temporomandibular joint disorders;
* The patient had an uncontrolled and/or untreated mental illness (e.g., severe depression and schizophrenia) for at least 6 months prior to the screening visit; Patients with a history of psychosis and/or mania within 5 years before screening were excluded;
* The patient has any other medical condition whose treatment takes precedence over MOH treatment or may interfere with the study treatment or impair compliance with treatment;
* Taking/using medications/stimulation devices that may affect headache (e.g., beta-blockers (atenolol, propranolol, metoprolol, etc.) due to headache or other reasons within 3 months before or during the screening period; Calcium channel blockers (flunarizine, benzothiazide, etc.); Antidepressants (amitriptyline, venlafaxine, duloxetine, etc.); Antiepileptic drugs (topiramate, sodium valproate, carbamazepine, etc); Angiotensin-receptor blockers (candesartan and lisinopril); Botulinum toxin; Gabapentin; Noninvasive vagus nerve stimulation, transcranial magnetic stimulation, peripheral trigeminal nerve stimulation; Biofeedback, health products; Occipital nerve block, other nerve block; Continuous infusion therapy, steroid reduction; Chiropractic therapy, physical therapy); Or treatment with injections (trigger point injections, extracranial nerve blocks or facet joint injections) on the head, face or neck;
* The patient has a history of moderate or severe head or neck trauma, or other neurological or systemic diseases (such as epilepsy and dementia) that the researcher believes may affect the central nervous system function;
* Patients have or have had one or more of the following conditions that were considered in the study to be associated with clinical symptoms: other neurological, pulmonary, hepatic, endocrine, gastrointestinal, hematologic, infectious, immunologic, or ocular conditions;
* A history of substance or alcohol abuse (according to DSM-5® criteria) within 24 months prior to the screening visit;
* During the screening or baseline visit, the patient has significant suicide risk (answers "Yes" to question 4 or 5 on the C-SSRS suicide ideation section, or answers "Yes" to any question regarding suicidal behavior at any time during the study on the C-SSRS);
* Prophylactic treatment for headache was received 1 month before the screening visit;
* One month before the screening visit, the patient had participated in a clinical study; Or had taken any medication for headache within the 5 plasma half-lives, whichever was longer, before the screening visit;
* Severe uncontrolled disease such as cancer, uncontrolled cardiovascular disease, severe hepatic and renal insufficiency, or coagulopathy; Women who are pregnant or preparing to become pregnant;
* Having known fear of acupuncture or having received acupuncture treatment within 8 weeks before enrollment;
* In the judgment of the investigators, the patients have diseases or take drugs that may affect the assessment of the safety, tolerability, or efficacy of the trial, or affect the conduct or interpretation of the study.
* Any one of the above items is excluded.

Inclusion Criteria for Patients with episodic migraine(Control group 1):

* According to the ICHD-3 criteria, it met the diagnostic criteria of episodic migraine; With/without tension-type headache;
* Headache days/month ≤6 days at enrollment;
* The number of days/month of using analgesics at enrollment was ≤6 days;
* Age between 18 and 80 years;
* Be able to fill out a headache diary;
* No previous history of drug abuse;
* No obvious comorbidities pain, physical or mental disorders;
* No alcohol or drug addiction;
* No pregnancy, breastfeeding, or plans for pregnancy in the next 12 months;

Inclusion Criteria for Healthy Participants(Control group 2):

* No headache or headache ≤2 days in the past 12 months at enrollment;
* No more than 6 days/month of use of analgesics at enrollment;
* Age between 18 and 80 years;
* No significant comorbidities pain, physical, or mental disorders;
* No organic, functional changes or systemic diseases that could cause headache;
* No history of head or neck trauma;
* No significant abnormalities in blood routine, biochemical tests, coagulation function, or urine routine in the past 12 months prior to enrollment;
* No alcohol or drug addiction;
* No pregnancy, breastfeeding, or plans for pregnancy in the next 12 months.

Nonrandomized patients with MOH:

●Participants who meet the MOH diagnostic criteria and fulfill the inclusion/exclusion criteria but decline randomization will be assigned to the non-randomized electroacupuncture group. These participants will receive electroacupuncture treatment directly, with no restrictions on the number of participants per center.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in the number of headache days | At the end of week 12 after randomization.
  Change from baseline in headache days per month

SECONDARY OUTCOMES:
Change in the number of headache days | At the end of week 4, week 8 after randomization; at week 24, week 36 of the follow-up period,
  Change from baseline in headache days per month
The proportion of responders | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The proportion of patients with at least a 50% reduction from baseline in headache days per month and no overuse of acute pain medications
The proportion of patients with at least 50% reduction in headache days per month | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The proportion of patients with at least 50% reduction in headache days per month from baseline
Change in mean daily headache duration | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The changes from baseline in mean daily headache duration
The proportion of patients with at least 50% reduction in mean daily headache duration | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The proportion of patients with at least 50% reduction in mean daily headache duration from baseline
Change in headache severity score per month | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The changes from baseline in headache severity score per month.
  Headache severity is recorded daily on a 0-3 scale:
  0 = No pain, 1 = Mild pain (does not interfere with activities), 2 = Moderate pain (interferes with some but not all activities), 3 = Severe pain (stops all activities) The monthly headache severity is calculated as the sum of the highest daily headache severity for each day in that month.
The proportion of patients with at least 50% reduction in headache severity score per month | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The proportion of patients with at least 50% reduction in headache severity score per month from baseline.
  Headache severity is recorded daily on a 0-3 scale:
  0 = No pain, 1 = Mild pain (does not interfere with activities), 2 = Moderate pain (interferes with some but not all activities), 3 = Severe pain (stops all activities) The monthly headache severity is calculated as the sum of the highest daily headache severity for each day in that month.
Change in the number of moderate and severe headache days per month | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The changes from baseline in the number of moderate and severe headache days per month
The proportion of patients with at least 50% reduction in the number of moderate and severe headache days per month | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The proportion of patients with at least 50% reduction in the number of moderate and severe headache days per month
Change in mean daily duration of moderate and severe headache | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The changes from baseline in mean daily duration of moderate and severe headache
The proportion of patients with at least 50% reduction in mean daily duration of moderate and severe headache | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The proportion of patients with at least 50% reduction in mean daily duration of moderate and severe headache
Change in number of days per month with acute medication for headache | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The changes from baseline in number of days per month with acute medication for headache
The proportion of patients with at least 50% reduction in number of days per month with acute medication for headache | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The proportion of patients with at least 50% reduction in number of days per month with acute medication for headache
Change in total number of doses taken per month for headache | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The changes from baseline in total number of doses taken per month for headache
The proportion of patients with at least 50% reduction in total number of doses taken per month for headache | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The proportion of patients with at least 50% reduction in total number of doses taken per month for headache
Change in Severity of Dependence Scale (SDS) | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The changes from baseline in the scores of Severity of Dependence Scale (SDS). The original SDS consists of five items, each scored on a scale from 0 to 3. A score of 0 indicates "never or almost never," whereas a score of 3 indicates "always or almost always." The psychological dependence score is based on the first four items of the SDS, with a maximum possible score of 12, higher scores indicate a greater level of dependence. The fifth item concerns the treatment process and is not related to the baseline.
Change in Hospital Anxiety and Depression Scale (HADS) | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The changes from baseline in the scores of Hospital Anxiety and Depression Scale (HADS).
  The HADS is used to assess anxiety and depression symptoms experienced over the past week. It consists of 14 items divided into two subscales (7 items each for anxiety and depression), with each item scored from 0 (no symptom) to 3 (severe symptom). Each subscale has a maximum score of 21, and higher scores indicate more severe symptoms. A score of ≥8 is defined as the presence of depression or anxiety.
Change in Headache Impact Test (HIT-6) | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The changes from baseline in the scores of Headache Impact Test (HIT-6). The HIT-6 is a brief tool for assessing the impact of headaches in clinical research and practice. It covers multiple domains of health-related quality of life, including pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. Each of the six items is rated on a 5-point Likert scale (6 = Never, 8 = Rarely, 10 = Sometimes, 11 = Very Often, 13 = Always). The total HIT-6 score is the sum of these six item scores and ranges from 36 to 78. Higher scores indicate a greater impact of headaches.
Change in Patient Global Impression of Change (PGIC) | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The changes in the scores of The Patient Global Impression of Change (PGIC). The PGIC is used to assess the participant's subjective evaluation of overall improvement. The scale consists of seven levels:1 = Very much improved, 2 = Much improved, 3 = Somewhat improved, 4 = No change, 5 = Somewhat worse 6 = Much worse, 7 = Very much worse. Lower scores indicate greater improvement.
Change in five-level version of EQ-5D (EQOL-5D-5L) | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  The changes from baseline in the five-level version of EQ-5D (EQOL-5D-5L).
  The EQ-5D-5L comprises two parts:
  1.EQ-5D Descriptive System:
  This system measures health status across five dimensions: Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression. Each dimension has five levels, rated from 1 to 5:
  1 = No problems/difficulty/discomfort, 2 = Slight problems/difficulty/discomfort 3 = Moderate problems/difficulty/discomfort, 4 = Severe problems/difficulty/discomfort, 5 = Extreme problems/difficulty/discomfort 2.EQ-5D Visual Analog Scale (VAS): This is a 20 cm vertical scale ranging from 0 to 100: 0 represents the "worst imaginable health", 100 represents the "best imaginable health". Higher scores on the VAS indicate better overall health status.
  This study uses the validated Chinese version of the EQ-5D-5L, which has demonstrated good reliability and validity.
Patients'expectation of the acupuncture efficacy | At baseline
  Participants are asked, "Do you think your medication overuse headache (MOH) improved after completing acupuncture treatment?" They select one of the following five responses: 1.Significantly improved, 2.Very much improved, 3.Some improvement, 4.No improvement at all, 5.Unclear.
  Lower-number responses (1 or 2) reflect greater perceived improvement compared with higher-number responses.
The patient blinding assessment | Within 5 minutes after the completion of any week 12 treatment session
  participants are informed that there are two acupuncture therapies: conventional electroacupuncture and micro-electroacupuncture. Both therapies are effective, and in both cases, participants may or may not feel electrical stimulation. They are then asked whether they would accept conventional electroacupuncture. The answer options are: Difficult to distinguish Yes No

OTHER OUTCOMES:
The proportion of patients with < 15 headache days per month | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
The proportion of patients with headache free days per month | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
The proportion of patients with cured Medication Overuse Headache(MOH) | At the end of week 4, week 8 and week 12 after randomization; at week 24, week 36 of the follow-up period,
  MOH-cured patients are those who no longer meet the criteria for MOH, with the following three conditions present:
  i) no acute medication overuse and remission of episodic headache; ii) no acute medication overuse, although chronic headache (≥15 headache days/month) remains,; iii) episodic headache, despite persistent medication overuse
The recurrence rate in patients with cured MOH | At week 24, week 36 of the follow-up period
  The recurrence rate is the proportion of individuals diagnosed with MOH at the end of follow-up among subjects who successfully abstinent
Brain MRI Data Analysis | At baseline and week 12 after randomization
  Evaluate the changes in the descending pain modulatory system in participants at baseline and after 12 weeks of treatment, including the gray matter structural covariance network, resting-state functional connectivity network, and deterministic tracking network of white matter fiber tracts.
  Randomly select 40 MOH patients (20 in the EA group and 20 in the SEA group) and 40 control group (20 in control group 1 and 20 in control group 2) for MRI scans. All participants from both the control group and the MOH patients are right-handed (i.e., habitually using their right hand for tasks such as writing, using chopsticks, and performing Fine motor skills), and the MRI scans must be conducted on the same model of machine.
Single-Cell Omics Outcome Analysis | 1.EA group: At baseline and week 12 after randomization; 2.SEA group: at week 12 after randomization.
  Single-Cell Omics and Phenotypic Changes in MOH Patients Versus healthy participants(control group 2).
  Blood samples are being collected from 6 MOH patients (3 from the EA group and 3 from the SEA group) and 3 healthy participants for single-cell transcriptome sequencing and analysis. All blood samples from both the control group and patients are collected at the same time of year.
Proteomic Outcome Analysis | At baseline and week 12 after randomization
  Proteomic and Phenotypic Changes in MOH Patients Versus healthy participants(control group 2) Blood samples are being collected from 30 MOH patients for proteomic testing and analysis. All blood samples from both the control group and patients are collected at the same time of year.
Metabolomics Outcome Analysis | At baseline and week 12 after randomization
  Metabolomics and Phenotypic Changes in MOH Patients Versus healthy participants(control group 2) Blood samples are being collected from 30 MOH patients for Metabolomics testing and analysis. All blood samples from both the control group and patients are collected at the same time of year.
Change in mean daily headache duration | At week 60, week 108 and week 156 of the follow-up period.
  The changes from baseline in mean daily headache duration
Change in mean daily duration of moderate and severe headache | At week 60, week 108 and week 156 of the follow-up period.
  The changes from baseline in mean daily duration of moderate and severe headache
Change in total number of doses taken per month for headache | At week 60, week 108 and week 156 of the follow-up period.
  The changes from baseline in total number of doses taken per month for headache
Change in number of days per month with acute medication for headache | At week 60, week 108 and week 156 of the follow-up period.
  The changes from baseline in number of days per month with acute medication for headache
The recurrence rate in patients with cured MOH | At week 60, week 108 and week 156 of the follow-up period.
  The recurrence rate is the proportion of individuals diagnosed with MOH at the end of follow-up among subjects who successfully abstinent
Change in Severity of Dependence Scale (SDS) | At week 60, week 108 and week 156 of the follow-up period.
  The changes from baseline in the scores of Severity of Dependence Scale (SDS) The original SDS consists of five items, each scored on a scale from 0 to 3. A score of 0 indicates "never or almost never," whereas a score of 3 indicates "always or almost always." The psychological dependence score is based on the first four items of the SDS, with a maximum possible score of 12, higher scores indicate a greater level of dependence. The fifth item concerns the treatment process and is not related to the baseline.
Change in Hospital Anxiety and Depression Scale (HADS) | At week 60, week 108 and week 156 of the follow-up period.
  The changes from baseline in the scores of Hospital Anxiety and Depression Scale (HADS) The HADS is used to assess anxiety and depression symptoms experienced over the past week. It consists of 14 items divided into two subscales (7 items each for anxiety and depression), with each item scored from 0 (no symptom) to 3 (severe symptom). Each subscale has a maximum score of 21, and higher scores indicate more severe symptoms. A score of ≥8 is defined as the presence of depression or anxiety.
Change in Headache Impact Test (HIT-6) | At week 60, week 108 and week 156 of the follow-up period.
  The changes from baseline in the scores of Headache Impact Test (HIT-6). The HIT-6 is a brief tool for assessing the impact of headaches in clinical research and practice. It covers multiple domains of health-related quality of life, including pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. Each of the six items is rated on a 5-point Likert scale (6 = Never, 8 = Rarely, 10 = Sometimes, 11 = Very Often, 13 = Always). The total HIT-6 score is the sum of these six item scores and ranges from 36 to 78. Higher scores indicate a greater impact of headaches.
Change in Patient Global Impression of Change (PGIC) | At week 60, week 108 and week 156 of the follow-up period.
  The changes in the scores of The Patient Global Impression of Change (PGIC). The PGIC is used to assess the participant's subjective evaluation of overall improvement. The scale consists of seven levels:1 = Very much improved, 2 = Much improved, 3 = Somewhat improved, 4 = No change, 5 = Somewhat worse 6 = Much worse, 7 = Very much worse. Lower scores indicate greater improvement.
Change in five-level version of EQ-5D (EQOL-5D-5L) | At week 60, week 108 and week 156 of the follow-up period.
  The changes from baseline in the five-level version of EQ-5D (EQOL-5D-5L).
  The EQ-5D-5L comprises two parts:
  1.EQ-5D Descriptive System:
  This system measures health status across five dimensions: Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression. Each dimension has five levels, rated from 1 to 5:
  1 = No problems/difficulty/discomfort, 2 = Slight problems/difficulty/discomfort 3 = Moderate problems/difficulty/discomfort, 4 = Severe problems/difficulty/discomfort, 5 = Extreme problems/difficulty/discomfort 2.EQ-5D Visual Analog Scale (VAS): This is a 20 cm vertical scale ranging from 0 to 100: 0 represents the "worst imaginable health", 100 represents the "best imaginable health". Higher scores on the VAS indicate better overall health status.
  This study uses the validated Chinese version of the EQ-5D-5L, which has demonstrated good reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Wang, Ph.D, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Department of Acupuncture and Moxibustion, China Academy of Chinese Medical Sciences Guang´anmen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data are available on reasonable request. You can send e-mail to us if you have any question
Supporting Information: Study Protocol, SAP
Time Frame: It depends
Access Criteria: It depends